CLINICAL TRIAL: NCT05685953
Title: A Randomized, Placebo-controlled, Double-blinded Phase I Study to Evaluate Safety and Immunogenicity of DNA Vaccine OC-007 as a Booster Dose of COVID-19 Vaccine
Brief Title: A Randomized, Phase I Study of DNA Vaccine OC-007 as a Booster Dose of COVID-19 Vaccine
Acronym: OpenCorona1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matti Sällberg (Other)
Responsible Party: Sponsor-Investigator, Matti Sällberg, Study Sponsor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Open Corona 1
Record Dates: First submitted 2023-01-11; First posted 2023-01-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Respiratory Infection; COVID-19 Vaccine Adverse Reaction
Keywords: Covid-19; DNA vaccine; booster dose; in vivo electroporation; adverse reactions; antibody levels; cellular immune response
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded phase I study including three dose levels of the DNA vaccine OC-007.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinding: subjects, study personnel and outcome assessors are blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active vaccine (Experimental): Plasmid DNA vaccine, OC-007
  Interventions: Biological: DNA vaccine OC-007
- Placebo (Placebo Comparator): Sodium chloride solution (0.9 %)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: DNA vaccine OC-007 — Plasmid DNA vaccine
  Other Names: COVID-19 vaccine
  Arms: Active vaccine
Other: Placebo — 0.9% NaCl solution
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blinded phase I study, designed to evaluate the safety including reactogenicity and immunogenicity of this investigational DNA vaccine delivered intramuscularly by in vivo EP in human adults. The vaccine doses will be given to healthy adults aged 18 to 60 years, who have been previously vaccinated against COVID-19 with 3 doses of either Comirnaty® or Spikevax®, or both in any combination ≥3 months ago.

DETAILED DESCRIPTION:
One dose of the investigational vaccine or placebo will be given as a fourth booster dose. The vaccine will be administered intramuscularly at 3 dose levels or given as placebo (containing a 0.9 % NaCl solution), in combination with in vivo EP. The EP method used in the study is a class IIa "EPS Gun" from IGEA optimized for Electro Gene Transfer (EGT) vaccination and CE marked for the intended use in this clinical trial.

Primary objective:

• The primary objective of this study is to assess the safety and reactogenicity of the investigational vaccine OC-007 DNA delivered by in vivo EP, as a booster dose given at ≥ 3 months post-initial mRNA vaccination.

The secondary objectives:

• To investigate the humoral immune response to the investigational vaccine administered as one dose, by measuring changes in spike and of nucleocapsid antibody levels.

Exploratory objective:

* To investigate in more detail the humoral response and analyze the cellular immune response to the investigational vaccine
* To evaluate the number of SARS-CoV-2 infections documented by positive PCR test during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 60 years (at the time of consent).
2. All study subjects have received three doses of registered mRNA vaccine/s, the last dose given ≥ 3 months before inclusion in this study.
3. Healthy participant, according to the investigator's clinical judgment, as established by medical history, vital signs, physical examination, and laboratory assessments.
4. No clinically significant laboratory abnormalities as determined by the investigator at screening.

   Note: one retest of lab tests is allowed within the screening window.
5. Negative HIV 1/2 antibody/antigen test, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody at screening.
6. Participant with a body mass index (BMI) 20-30.0 kg/m2.
7. Provide written informed consent before initiation of any study procedures.
8. A female participant is eligible for this study if she is one of the following:

   * of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year)
   * of childbearing potential but agrees to practice highly effective contraception or abstinence (if this is the preferred and usual lifestyle of the participant) from 30 days prior to vaccination up to 3 months after vaccination.

   Highly effective methods of contraception include one or more of the following:
   1. male partner who is sterile (vasectomised) prior to the female study subject's entry into the study and is the sole sexual partner for the female subject;
   2. hormonal (oral, intravaginal, transdermal, implantable or injectable)
   3. an intrauterine hormone-releasing system (IUS)
   4. an intrauterine device (IUD) with a documented failure rate of < 1%.
9. A female participant is eligible if she is willing to abstain from donating oocyte from the screening visit up to 3 months after vaccination.
10. A male participant who is sexually active is eligible if he is willing to use a condom from the screening visit up to 3 months after vaccination except if the male participant is sterile (e.g. vasectomised); the unique female sexual partner is postmenopausal, is permanently sterilized (e.g. hysterectomy or tubal ligation), or use a highly effective method of contraception.
11. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study.

Exclusion Criteria:

1. Previous vaccination with investigational or registered non-mRNA vaccines against COVID-19.
2. History of presence of pulmonary disorders (chronic obstructive pulmonary lung disease etc) or asthma (exception of allergic asthma, which is allowed).
3. History or presence of thrombocytopenia and/or bleeding disorders.
4. A positive serum pregnancy test at screening or urine pregnancy test prior to study injection, women who are planning to become pregnant during the study, or women who are breastfeeding.
5. Clinically relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, inflammatory, autoimmune, central nervous system or neurological diseases.
6. Use of immunosuppressive drugs as e.g. corticosteroids (excluding topical preparations and inhalers) within 3 months prior to vaccination or 6 months for chemotherapies and all along the study.
7. Vaccination within 2 weeks prior to vaccination or planning to receive a licensed vaccine before month 3 (e.g. inactivated influenza vaccine).
8. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of known or suspected allergic reaction likely to be exacerbated by any component of the Investigational vaccine.
9. Participation in another investigational clinical study within four weeks before the screening visit or planned before the study completion.
10. Subjects with confirmed or suspected immunodeficiency.
11. SARS-CoV-2 infection within the past 2 weeks3 months prior to enrolment, or ongoing symptom of COVID-19.
12. Any condition that in the opinion of the principal investigator (PI) would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Local reactions after the vaccine/placebo dose | Up to 7 days after the vaccine/placebo dose
  Local reactions (pain at the injection site, redness, and swelling) for up to 7 days after the vaccine/placebo dose
Visual analogue scale pain rating scale score | At 0, 5, 15, 30 and 60 minutes post-EP.
  Visual analogue scale (VAS) score to rate the level of pain experienced immediately (0 minutes), and after 5, 15, 30 and 60 minutes post-EP. Scale is continous and the farther right on the scale line the more pain.
Systemic events for 7 days after each vaccine/placebo dose. | For 7 days after each vaccine/placebo dose.
  Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain) for 7 days after each vaccine/placebo dose.
Unsolicited AEs | From the study dose to 28 days after vaccination.
  Unsolicited AEs from the study dose to 28 days after vaccination.
Serious Adverse Events (SAEs)/SUSARs | From the study dose until the study end at 3 months after vaccination.
  Serious Adverse Events (SAEs)/suspected unexpected serious adverse reactions (SUSARs) from the study dose until the study end at 3 months after vaccination.

SECONDARY OUTCOMES:
Change from baseline in antibody levels to the SARS-CoV-2 spike and nucleocapsid protein. | Day 7, Day 14, 1 Month and 3 Months.
  Change from baseline sample (a two-fold increase in endpoint titer or a 50% increase in optical density at a 1:62, 1:125, 1:250, 1:500, or 1:1000 serum dilution) in antibody levels to the SARS-CoV-2 spike and nucleocapsid protein by inhouse and/or commercial assays during the study period.

OTHER OUTCOMES:
Exploratory: In depth humoral and cellular immunological responses | Day 7, Day 14, 1 Month and 3 Months
  Description of in depth humoral and cellular immunological responses after receiving investigational vaccine at each sampling. Immunoglobulin levels analysed by Enzyme-Linked Immunosorbent Assays (ELISAs). Antibody titer analysed by CPE based microneutralization assay. Isolated Peripheral Blood Mononuclear Cell behavior analysed by enzyme-linked immunospot (ELISpot) assay. Flow cytometry will be used for functional and phenotypic characterization of T-cells.
Exploratory: SARS-CoV-2 infections | Up to 3 Months
  Number and severity of SARS-CoV-2 infections during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Sällberg, PhD, Study Director — Department of Laboratory Medicine, Karolinska Institute, Stockholm
Locations (1):
- Phase I Study Unit, Karolinska University Hospital, Stockholm, Region Stockholm, Sweden